CLINICAL TRIAL: NCT04911725
Title: Study of the Effect of an Elastic Compression Medical Device (Prototype), on Water Balance Change in Healthy Subjects. Exploratory, Randomized, Open-label, Controlled and Crossover Study
Brief Title: Study of the Effect of an Elastic Compression Medical Device, on Water Balance Change in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Innothera (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CVE101-17
Record Dates: First submitted 2021-05-19; First posted 2021-06-03 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome (OSAHS)
Keywords: OSAHS; Elastic compression device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With device use (Experimental): Volunteers included will use IMD during one of the two periods of the study.
  Interventions: Device: Elastic Compression Prototype
- Without device use (No Intervention): Volunteers included will not use IMD during the other period of the study (reverse of experimental)

INTERVENTIONS:
Device: Elastic Compression Prototype — Elastic Compression device - No medical, surgical or laboratory procedure is implied in the use of the IMD.
  Arms: With device use

SUMMARY:
Obstructive sleep apnea-hypopnea syndrome (OSAHS) is characterized by the occurrence of abnormally frequent episodes of interrupted ventilation (apnea) or significant reduction of ventilation (hypopnea) during sleep. It is linked to a repeated collapse of the upper airways during sleep.

Episodes of apnea and hypopnea cause hypoxemia and micro-awakenings with a well-established impact on quality of life and daily activities. Physiologically, OSAHS can be aggravated when moving from a standing to a supine position through fluid shift from the lower limbs to the upper body, thereby modifying the opening of the upper airways. A decrease of the water balance by bilateral diurnal compression of the lower limbs (during daytime in standing position) may limit this nocturnal fluid shift (at night in supine position) and thus reduce the severity of OSAHS.

Two comparative clinical trials [Redolfi 2011; White 2015] have shown a clinically modest reduction of sleep apnea (-36% and -27%, respectively), which was however statistically significant versus untreated control group (p = 0.002 and p = 0.04, respectively), when elastic compression medical devices of 20 to 30 mmHg were worn during the daytime. The hypothesis of fluid shift influence on OSAHS has been tested [Berg 1993; Redolfi 2011; White 2015], but the decrease of the water balance when the device is used remains to be quantified.

The CVE101-15 exploratory clinical investigation sponsored by Laboratoires Innothera performed on healthy volunteers confirmed the hypothesis of a diuretic effect of elastic compression stockings applying a pressure of 33 mmHg at the ankle, worn for 13-14 hours during the daytime for 3 days, with a good safety profile of this device. Moreover, it enabled the identification of reliable parameters and the endpoints to be used to demonstrate a diuretic effect.

Based on this information, there may be a real interest in conducting further investigations about the evolution of water balance beyond a 3-day period of elastic compression use in the daytime.

Hence, the main objective of this clinical investigation is to compare precisely, under standardized test conditions, water balance changes in healthy subjects over 5 days with or without daytime use of the investigational medical device (IMD), an elastic compression device prototype specially designed for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject aged 40 years old or more.
2. Subject with a body mass index (BMI) between 18.5 and 30 kg/m².
3. Healthy subject, registered in the French biomedical research volunteer national file.
4. Subject for whom both lower limb measurements correspond to the size grid of the IMD used.
5. Subject agreeing to abstain from alcohol intake from 48 hours before P1D-2, during all hospitalization periods and during the outpatient period.
6. Subject accepting to proceed with a COVID-19 test at the time of each inpatient period, and for whom the result is negative
7. Subject accepting to protect himself in an appropriate way to avoid COVID-19 infection during the outpatient period.
8. Subject practicing under 5 hours of intense physical activity per week, on average, in the 4 weeks preceding the screening visit (e.g. no marathon training or military training).
9. Subject agreeing to abstain from any strenuous activity, especially sports, from the screening visit to the end of clinical investigation (including during the outpatient period).
10. Subject accepting the constraints of the clinical investigation.
11. Subject being available for the duration of the clinical investigation.
12. Subject who has signed the informed consent form (ICF) after being adequately informed and receiving the information sheet.
13. Subject affiliated with the French social security system or receiving benefits of that type.

Exclusion Criteria (non-inclusion criteria):

1. Subject who is a smoker or a former smoker who stopped smoking less than 6 months ago.
2. Subject following a salt-free diet.
3. Subject following or planning to follow either a slimming diet or any specific diet that could not be followed during hospitalization.
4. Subject having a temperature > 38.0°C at screening or in the morning of D-2 and D1 of the first period (P1).
5. Subject having, upon clinical examination, an abnormal systolic blood pressure (SBP), diastolic blood pressure (DBP) or heart rate (HR) judged clinically significant by the Investigator.
6. Subject having an intestinal transit disorder that disrupts hydroelectric balance.
7. Alcohol-dependent subject or subject with a positive alcohol breath test.
8. Subject having a localized or general edema (a simple evening edema of the legs or ankles is accepted for inclusion).
9. Subject suffering from insulin-dependent or uncontrolled diabetes (controlled diabetes is accepted).
10. Subject with a serious, stabilized, or progressive illness (as judged by the Investigator).
11. Subject with hypertension or heart failure.
12. Subject with known renal function disorders.
13. Subject with known liver failure.
14. Subject with venous insufficiency of clinical class C3, C4, C5 or C6 according to the Clinical / Etiological / Anatomical / Pathophysiological (CEAP) classification.
15. Subject having a medical background of deep and superficial vein thrombosis.
16. Subject following long-term therapy with diuretics, nonsteroidal anti-inflammatory drugs (NSAIDs), steroids, nutritional supplements or opiates.
17. Subject having, upon questioning or clinical examination, advanced peripheral neuropathy, skin infections, eczematous dermatitis, or weeping skin disorder of the legs.
18. Subject with a medical contraindication to compression therapy according to the interview or clinical examination: phlegmatia coerulea dolens, septic thrombosis, intolerance to the IMD, allergic reaction to any component, arteritis obliterans of lower limbs, advanced diabetic microangiopathy.
19. Subject with active implants, such as a pacemaker or artificial heart type, and non-active implants, for example a hip prosthesis (dental implants are authorized).
20. Subject who is participating in another clinical trial or who is in the exclusion period from a previous study/clinical investigation.
21. Person deprived of freedom by judicial or administrative decision, or a person hospitalized without his consent.
22. Subject of legal age who is protected by law or under guardianship.
23. Subject with a current mental or psychiatric disorder or a history of mental or psychiatric disorder, or any other factor limiting the collection of informed consent.
24. Person who works for the CRO or for Laboratoires Innothera, or has a dependent relationship with these entities.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
EFFICACY: Compare the cumulative evolution of the water balance over a period of 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine (24h sequence), with or without daytime use of the IMD | 5 consecutive days
  Cumulative evolution of the water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.

SECONDARY OUTCOMES:
EFFICACY: Compare the mean daily water balance estimated over a period of 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine every day during 5 days, with or without daytime use of the IMD | 5 days
  Mean daily water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.
EFFICACY: Compare the cumulative evolution of the daytime water balance over 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine during the daytime sequence, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the daytime water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.
EFFICACY: Compare the mean daily daytime water balance estimated over 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine during the daytime sequence, with or without daytime use of the IMD | 5 days
  Mean daily daytime water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.
EFFICACY: Compare the cumulative evolution of the nighttime water balance over 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine during the nighttime sequence, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the nighttime water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.
EFFICACY: Compare the mean daily nighttime water balance estimated over 5 days, assessed by the adjusted difference between the volume of fluid intake and the volume of urine during the nighttime sequence, with or without daytime use of the IMD | 5 days
  Mean daily nighttime water balance over a period of 5 days, assessed by the difference between the volume of fluid intake, determined by weight, and the volume of the urine, determined by weight, with or without daytime use of the IMD.
EFFICACY: Compare the cumulative evolution of the subject's weight over 5 days, assessed by the adjusted difference between the weight at the end of the 5-day period and the weight at the start of the 5-day period, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily subject's weight evolution estimated over 5 days, assessed by the adjusted difference between the weight at H0 and the weight at H0 the following day, with or without daytime use of the IMD | 5 days
  Mean daily evolution of the subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the daytime subject's weight over a period of 5 days, assessed by the adjusted cumulative differences between the weight between H0 and H14 each day, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the daytime subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily daytime subject's weight evolution estimated over a period of 5 days, assessed by the adjusted difference between the weight at H0 and the weight at H14 each day, with or without daytime use of the IMD | 5 days
  Mean daily daytime evolution of the subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the nighttime subject's weight over 5 days, assessed by the adjusted cumulative differences between the weight between H14 and H0 of the following day each day, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the nighttime subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily nighttime subject's weight evolution estimated over 5 days, assessed by the adjusted difference between the weight at H14 and the weight at H0 of the following day each day, with or without daytime use of the IMD | 5 days
  Mean daily nighttime evolution of the subject's weight over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the urine volume over a period of 5 days, assessed by the adjusted cumulative volumes of urine, with or without daytime use of the IMD (24h sequence) | 5 days
  Cumulative evolution of the urine volume over a period of 5 days, with or without daytime use of the IMD
. EFFICACY: Compare the mean daily urine volume estimated over a period of 5 days, assessed by the adjusted daily volumes of urine, with or without daytime use of the IMD (24h sequence) | 5 days
  Mean daily urine volume over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative daytime evolution of the urine volume over a period of 5 days, assessed by the adjusted cumulative volumes of daytime urine, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the daytime urine volume over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily daytime urine volumes estimated over a period of 5 days, assessed by the adjusted daily daytime volumes of urine, with or without daytime use of the IMD | 5 days
  Mean daily daytime urine volume over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative nighttime evolution of the urine volume over a period of 5 days, assessed by the adjusted cumulative volumes of nighttime urine, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the nighttime urine volume over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily nighttime urine volumes estimated over a period of 5 days, assessed by the adjusted daily nighttime volumes of urine, with or without daytime use of the IMD | 5 days
  Mean daily nighttime urine volume over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative daily evolution of the neck circumference (dynamic and supine sequences) over a period of 5 days, with or without daytime use of the IMD (24h sequence) | 5 days
  Cumulative evolution of the daily neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily evolution of the neck circumference (dynamic and supine sequences) over a period of 5 days, with or without daytime use of the IMD (24h sequence) | 5 days
  Mean daily evolution of the neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the neck circumference in the dynamic sequence over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the dynamic sequence neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean dynamic sequence evolution of the neck circumference over a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean dynamic sequence evolution of the neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the neck circumference in the supine sequence over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the supine sequence neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean supine sequence evolution of the neck circumference over a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean supine sequence evolution of the neck circumference over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative daily evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thigh (dynamic and supine sequences) over 5 days, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the daily leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thigh (dynamic and supine sequences) over 5 days, with or without daytime use of the IMD | 5 days
  Mean daily evolution of the leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thigh in the dynamic sequence over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the dynamic sequence leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean dynamic sequence evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thighover a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean dynamic sequence evolution of the leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thigh in the supine sequence over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative evolution of the supine sequence leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean supine sequence evolution of the leg perimeters at 3 points, at the thinnest part of the ankle, at the largest part of the calf and at mid-thigh over a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean supine sequence evolution of the leg perimeters at 3 points over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative daily evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD (24h sequence) | 5 days
  Cumulative daily evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daily quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD (24h sequence) | 5 days
  Mean daily quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative daytime evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative daytime evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean daytime quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean daytime quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the cumulative nighttime evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD | 5 days
  Cumulative nighttime evolution of the quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
EFFICACY: Compare the mean nighttime quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD | 5 days
  Mean nighttime quantity of NaCl excreted in the urine over a period of 5 days, with or without daytime use of the IMD
ACCEPTABILITY: Describe the acceptability of the IMD during daytime use | 5 days
  Responses to acceptability questionnaire each day of IMD use
SAFETY: Describe the safety of the IMD use during daytime use | 5 days
  Emergent adverse events (EAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie HAYS, MD, Principal Investigator — Biotrial
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: No